CLINICAL TRIAL: NCT01483534
Title: Evaluation of the Innovative Pulmonary Solutions (IPS) System for Targeted Lung Denervation (TLD) Therapy in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) - A Safety Study
Brief Title: Innovative Pulmonary Solutions (IPS) System for Targeted Lung Denervation
Acronym: IPS-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvaira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-001
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; Pulmonary; Intervention; Device; Denervation; Lung; Holaira, Inc.; Innovative Pulmonary Solutions, Inc.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Targeted Lung Denervation (Experimental): Targeted Lung Denervation
  Interventions: Device: TLD Therapy (IPS SystemTM)

INTERVENTIONS:
Device: TLD Therapy (IPS SystemTM) — Targeted Lung Denervation Therapy will be achieved bronchoscopically. As this is a single-arm, non-randomized study, it is anticipated that all patients who provide written informed consent and meet the protocol entry criteria will undergo treatment.
  Other Names: TLD Therapy, Targeted Lung Denervation Therapy

SUMMARY:
The purpose of this study is to evaluate the safety of Targeted Lung Denervation Therapy (or TLD TherapyTM) in patients suffering from COPD. Technical feasibility of the IPS SystemTM will also be evaluated through confirmation of successful application of TLD Therapy.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 30% to 60%
* FEV1/FVC <70%
* Prior smoker (at least 10 pack years)
* Quit smoking for at least 6 months

Exclusion Criteria:

* Pulmonary hypertension, peripheral edema suggesting CHF or polycythemia
* Prior lung transplant, LVR, LVRS, median sternotomy, bullectomy or lobectomy
* Pulmonary nodule requiring surgery
* Presence of implantable electronic devices
* Active respiratory infection within recent weeks
* COPD exacerbation within recent weeks
* Recent Myocardial infarction (MI)
* Recent and unstable or life threatening arrhythmia
* Malignancy treated with radiation or chemotherapy within the last 2 years
* Presence or clinical diagnosis of other respiratory diseases other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 365 days post procedure
  Safety will be evaluated as freedom from documented and sustained worsening of COPD directly attributable to the investigational device or procedure.

SECONDARY OUTCOMES:
Technical Feasibility | At time of Treatment
  The ability to access the target treatment area and deliver RF energy to the target treatment site.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (3):
- University Medical Center Groningen (UMCG), Groningen, Netherlands
- South Africa (2):
  - Panorama Medi-Clinic, Panorama, Cape Town
  - Stellenbosch University, Capetown

REFERENCES:
- [Result] Slebos DJ, Klooster K, Koegelenberg CF, Theron J, Styen D, Valipour A, Mayse M, Bolliger CT. Targeted lung denervation for moderate to severe COPD: a pilot study. Thorax. 2015 May;70(5):411-9. doi: 10.1136/thoraxjnl-2014-206146. Epub 2015 Mar 4. PMID 25739911
- See also: Targeted lung denervation for moderate to severe COPD: a pilot study. — http://thorax.bmj.com/content/early/2015/03/03/thoraxjnl-2014-206146